CLINICAL TRIAL: NCT02478567
Title: The Effect of Axioscapular and Rotator Cuff Exercise Training Sequence in Patients With Subacromial Impingement Syndrome: A Randomized Crossover Trial
Brief Title: Exercise Training Sequence for Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ed Mulligan, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 052012-017
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Scapular Training (Experimental): Initiated scapular training exercise for the first 4 weeks followed by addition of rotator cuff exercises the next four weeks
  Interventions: Other: Scapular Training
- Rotator Cuff Training (Experimental): initiated rotator cuff training exercise for the first 4 weeks followed by addition of scapular training exercises the next four weeks.
  Interventions: Other: Rotator Cuff Training

INTERVENTIONS:
Other: Rotator Cuff Training — four specific band-resisted strength training exercises for scapula
  Other Names: exercise
  Arms: Rotator Cuff Training
Other: Scapular Training — four specific band-resisted strength training exercises for rotator cuff
  Other Names: exercise
  Arms: Scapular Training

SUMMARY:
Randomized crossover trial evaluating the impact of exercise training sequence of axioscapular and rotator cuff exercises in patients diagnosed with subacromial impingement syndrome.

DETAILED DESCRIPTION:
While physical therapy is an effective element in the rehabilitation of rotator cuff (RC) disease, the most effective sequence of training interventions has not been defined. The purpose of this study is to determine if there is a difference in pain or function in patients who are given RC strengthening prior to or after initiating scapular stabilization exercises.

The study was a prospective randomized crossover design. 26 men and 14 women, mean age 51, diagnosed with subacromial impingement syndrome (SAIS) were randomly assigned to one of two groups for a comprehensive and standardized rehabilitation program over six visits at an orthopedic outpatient clinic. One group was prescribed a 4-week program of scapular stabilization exercises while the other group began with RC strengthening exercises. The crossover design had each group add the previously excluded four exercises to their second month of rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* diagnosis of Neer Stage I/II subacromial impingement with a primary pain complaint in the shoulder and/or upper arm
* presence of at least two of the following findings: painful arc, weakness in external rotation, positive impingement sign (Hawkins-Kennedy or Neer/Walsh tests), pain and/or weakness with resistance to internal rotation, external rotation, or scapular plane elevation.

Exclusion Criteria:

* concurrent medical co-morbidities including pregnancy, diabetes, and rheumatoid arthritis -
* osteoarthritis greater than grade 2 on the Kellgren-Lawrence scale
* current diagnosis and/or previous history of glenohumeral instability or dislocation
* full-thickness rotator cuff tear
* adhesive capsulitis
* fractures of the scapula, clavicle or humerus
* scapulothoracic or rotator cuff paresis
* shoulder surgery in past year
* inability to speak the English language at a level sufficient to obtain informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
American Shoulder Elbow Surgeon's Outcome Score | 16 weeks
  self-report of function
Numeric Pain Score | 16 weeks
  pain levels
Global Rating of Change | 16 weeks
  patient satisfaction
Global Percentage of Improvement | 16 weeks
  patient perception of status

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States